CLINICAL TRIAL: NCT04122950
Title: Exergaming to Increase Physical Activity in Overweight/Obese Children and Adolescents
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Few interested participants
Sponsor: Norwegian University of Science and Technology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2019/1082
Record Dates: First submitted 2019-09-30; First posted 2019-10-10 (Actual); Last update posted 2022-04-07 (Actual); Status verified 2022-03

CONDITIONS: Obesity
Keywords: Exercise therapy; Physical fitness; Gaming; Child; Healthy lifestyle; Fitness testing
MeSH Terms: conditions — Obesity | interventions — Exergaming

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exergaming (Experimental): The participants in the Exergaming group will use the PlayPulse exergame for 45 minutes a minimum of two times per week for 8 weeks. Between 8 and 12 weeks the exergaming group will be provided with free access to the exergame but without the two mandatory exergaming sessions
  Interventions: Behavioral: Exergaming
- Control (No Intervention): Continue with normal daily routine.

INTERVENTIONS:
Behavioral: Exergaming — The participants in the Exergaming group will use the PlayPulse exergame for 45 minutes a minimum of three times per week for 8 weeks. Between 8 and 12 weeks the exergaming group will be provided with free access to the exergame but without the two mandatory exergaming sessions
  Arms: Exergaming

SUMMARY:
The primary purpose of this study is to examine the effects of regular exergaming for 8 weeks in 24 overweight/obese children and adolescents (10-17 years) on maximal aerobic fitness (VO2max) and physical activity levels measured before and after (8 weeks) intervention period, and in addition at follow-up (12 weeks). We also wish to investigate the effects on markers of cardio metabolic health and body composition, measured at baseline, 8 weeks and 12 weeks follow-up.

Also, the participants gaming frequency will be registered throughout the 8 week period, as well as during the follow-up between 8 and 12 weeks. Aim of this study is to investigate if access to this game can provide health benefits for overweight/obese children and adolescents.

ELIGIBILITY:
Inclusion Criteria:

* Defined as overweight/obese for age and sex
* Able to ride a bike for up to 60 minutes

Exclusion Criteria:

* Known cardiovascular disease
* Taking beta-blockers or anti-arrhythmic drugs
* Other diseases that restrict them from doing High-Intensity Training

Ages: 10 Years to 24 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 6 (Actual)
Dates: Start 2020-02-24 (Actual); Primary Completion 2022-03-28 (Actual); Study Completion 2022-03-28 (Actual)

PRIMARY OUTCOMES:
Daily time physical activity (moderate, vigorous and very vigorous) | 12 weeks
  Measured by activity monitors (SenseWear Armband) which participants will wear for one week at start of intervention period and at 12 weeks.

SECONDARY OUTCOMES:
Daily average energy expenditure | 8 and 12 weeks
  Measured by activity monitors (SenseWear Armband) which participants will wear for one week at start of intervention period, 8 weeks and 12 weeks.
Daily average number of steps | 8 and 12 weeks
  Measured by activity monitors (SenseWear Armband) which participants will wear for one week at start of intervention period, 8 weeks and 12 weeks.
Daily time in sedentary activity (< 3.0 metabolic equivalents = METs) | 8 and 12 weeks
  Measured by activity monitors (SenseWear Armband) which participants will wear for one week at start of intervention period, 8 weeks and 12 weeks.
Daily time in moderate intensity activity (3.0-6.0 metabolic equivalents = METs) | 8 and 12 weeks
  Measured by activity monitors (SenseWear Armband) which participants will wear for one week at start of intervention period, 8 weeks and 12 weeks.
Daily time in vigorous intensity activity | 8 and 12 weeks
  Measured by activity monitors (SenseWear Armband) which participants will wear for one week at start of intervention period, 8 weeks and 12 weeks.
Daily time in very vigorous intensity activity (>9.0 metabolic equivalents = METs) | 8 and 12 weeks
  Measured by activity monitors (SenseWear Armband) which participants will wear for one week at start of intervention period, 8 weeks and 12 weeks.
Daily average total physical activity duration | 8 and 12 weeks
  Measured by activity monitors (SenseWear Armband) which participants will wear for one week at start of intervention period, 8 weeks and 12 weeks.
Bioelectrical impedance | 8 and 12 weeks
  Body composition assessed using bioelectrical impedance analysis (InBody 720)
Blood Pressure | 8 and 12 weeks
Fasting circulating glucose, as blood marker of cardiometabolic health | 8 and 12 weeks
Fasting triglycerides, LDL-, HDL- and Total cholesterol, as blood marker of cardiometabolic health | 8 and 12 weeks
Circulating insulin concentration, as blood marker of cardiometabolic health | 8 and 12 weeks
glucose response to a 2 hour glucose tolerance test, as blood marker of cardiometabolic health | 8 and 12 weeks
VO2max | 8 and 12 weeks
  Maximal Aerobic Capacity
Daily time physical activity (moderate, vigorous and very vigorous) | 8 weeks
  Measured by activity monitors (SenseWear Armband) which participants will wear for one week at start of intervention period and at 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Øystein Risa, Study Director — Norwegian University of Science and Technology; Trine Moholdt, PhD, Principal Investigator — Norwegian University of Science and Technology
Locations (1):
- Department of Circulation and Medical Imaging, Trondheim, Norway

IPD SHARING:
Plan to Share IPD: Undecided